CLINICAL TRIAL: NCT01210924
Title: Chinese Study of Pediatric Antiretroviral Therapy
Brief Title: Chinese Network of Pediatric Antiretroviral Therapy
Acronym: CN-PART
Status: Completed | Type: Observational
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Other Study IDs: Pediatric treatment 2010; 2008ZX10001-007 (Other Grant/Funding Number: Chinese Ministory of Health)
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2013-11

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: children; Acquired Immunodeficiency Syndrome; antiretroviral therapy; China; Mortality
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plamsa, PMBC, whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric ART patients

SUMMARY:
This is an observational cohort in pediatric HIV patients in China. Children who receive antiretroviral drugs will be recruited in this study. The main objectives are as follows: 1. To establish simpler and smarter pediatric antiretroviral therapy in China including both first-line and second-line regimens. 2. To study the nature, characteristics and mechanisms of immunoreconstitution in HIV-infected children using the data and samples from the pediatric antiretroviral therapy cohort. 3. To establish a basic science and clinical research network based on the pediatric antiretroviral cohort.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of HIV infection
* receiving triple antiretroviral drugs

Exclusion Criteria:

* clinical status not stable

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric HIV-infected patients receiving triple antiretroviral drugs
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The immunology and virologic outcomes | 2016

CONTACTS AND LOCATIONS:
Overall Officials: Fujie Zhang, MD, Principal Investigator — National Center for AIDS/STD control and prevention
Locations (1):
- National Center for AIDS/STD Control and Prevention, China Center for Disease Control and Prevention, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided